CLINICAL TRIAL: NCT00854971
Title: Evaluating the Safety and Efficacy of Combination Therapy With FOLFOX-4 and TKcell Therapy Versus FOLFOX-4 Alone in Patients With Recurrent, Unresectable and Advanced Colorectal Cancer
Brief Title: Efficacy Study of TKcell in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Binex (Industry)
Responsible Party: Park, Eun-Jin / Research institute, CRM(clinical research manager)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX-TK-002
Record Dates: First submitted 2009-02-28; First posted 2009-03-03 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-03

CONDITIONS: Advanced Colorectal Cancer
Keywords: NKCell; FOLFOX-4; advanced or unresectable colorectal cancer
MeSH Terms: interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Oxaliplatin infusion (85mg/m2) on days 1 and 15 (every 2 weeks) 5-FU bolus + infusions (400 mg/m2) on days 1, 2, 15 and 16 LV infusions (200 mg/m2) on days 1, 2, 15 and 16
- Active (Active Comparator): FOLFOX-4 regimen + Infusion of TKCell(autologous activated lymphocyte) over 2x10^9 cells, IV route, 7 times
  Interventions: Biological: TKCell

INTERVENTIONS:
Biological: TKCell — Biological/Vaccine: TKCell
  Other Names: NKCell; FOLFOX-4
  Arms: Active

SUMMARY:
The purpose of this study is to determine efficacy of NKCell in colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Diagnosis of histologically confirmed adenocarcinoma of the colorectal
* ECOG performance status of 0 - 2
* At least one definite measurable lesion(s): ≥ 1 cm on spiral CT scan or ≥2cm in physical examination
* Adequate liver, renal, bone marrow functions as evidence by the following;
* Absolute neutrophil count > 1.5 x 109/L; platelets > 7.5 x 109/L; Bilirubin less than 2 mg/dL ASAT and/or ALAT < 5 UNL; serum creatinine ≤ 2 ULN
* Minimum life expectancy of 12 weeks
* Effective contraception for both male and female subjects if the risk of conception exists

Exclusion Criteria:

* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Previous chemotherapy for gastric cancer except adjuvant treatment with progression of disease documented > 6 months after end of adjuvant treatment.
* Previous oxaliplatin-based chemotherapy
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to randomization and chemotherapy
* HIV antibody (+), Chronic hepatitis
* Uncontrolled infection
* Concurrent or previous chronic systemic immune therapy, targeted therapy, hormonal therapy not indicated in the study protocol except for contraception
* Clinically relevant coronary artery disease, history of myocardial infarction, high risk of uncontrolled arrhythmia
* Known hypersensitivity reaction to any of the components of the treatment.
* Pregnancy (absence to be confirmed by ß-hCG test) or lactation period
* Participation in another clinical study within the 30 days before randomization
* Significant disease which, in the investigator's opinion, would exclude the subject from the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Determine response rate | within study period

SECONDARY OUTCOMES:
Determine safety of combination,time to treatment failure, overall survival time | within study period

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Goo Cho, M.D, Ph.D, Principal Investigator — The Catholic Medical Center
Locations (1):
- The Catholic University of Korea, Seoul, Banpo-dong, South Korea

REFERENCES:
- See also: (Click here for more information about this study.) — http://www.bi-nex.com/